CLINICAL TRIAL: NCT06130657
Title: Volumetric Analysis of Maxillary Sinus After Guided Lateral Sinus Lift Procedure With Simultaneous Implant Placement
Brief Title: Volumetric Analysis of Maxillary Sinus After Guided Lateral Sinus Lift Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Zewail (Other)
Responsible Party: Sponsor-Investigator, Ahmed Zewail, Resident at the Department of Oral and Maxillofacial Surgery, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUAREC202100012-06
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Lateral Sinus Lifting; Dental Implant
Keywords: Sinus lifting; Dental implant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Lateral Maxillary Sinus Floor Elevation using surgical guide (Active Comparator)
  Interventions: Procedure: Lateral Maxillary Sinus Floor Elevation using surgical guide
- Group 2: Lateral Maxillary Sinus Floor Elevation without surgical guide (Active Comparator)
  Interventions: Procedure: Lateral Maxillary Sinus Floor Elevation without surgical guide

INTERVENTIONS:
Procedure: Lateral Maxillary Sinus Floor Elevation using surgical guide — The surgical procedure begins with securing a prefabricated guide firmly to the surgical site. Implant positions are marked, and after guide removal, a crestal incision is made 1 mm palatal to the marked point, extending with sulcular and vertical incisions. A full-thickness mucoperiosteal flap is reflected to expose the maxillary sinus and alveolar crest. After readapting the surgical guide to the bone, implant positions are marked, and cutting edges are tracked. The lateral window is formed by extending and connecting mesial and distal borders, created using piezotome. The sinus membrane is carefully reflected and elevated with a surgical curette to avoid iatrogenic perforation. Implant fixtures are then placed using the identical surgical guide, followed by graft material placement beneath the elevated sinus membrane. If the bony plate is preserved, the lateral window is covered with the plate.
  Arms: Group 1: Lateral Maxillary Sinus Floor Elevation using surgical guide
Procedure: Lateral Maxillary Sinus Floor Elevation without surgical guide — The sinus's lateral wall is exposed through a crestal incision and a mucoperiosteal flap. A bony window is created, and upon its removability, the sinus floor is carefully elevated using sinus elevation curettes, taking care to avoid membrane perforation. In cases of perforation, a resorbable collagen membrane is applied to cover the hole. Implant osteotomies are then completed following the standard sequential placement protocol. Graft material, mixed with normal saline, is gently packed into the sinus to fill the cavity with bone substitute material and achieve the desired bone height. Finally, a resorbable membrane is placed on the outer surface of the window, and the flap is sutured for primary closure.
  Arms: Group 2: Lateral Maxillary Sinus Floor Elevation without surgical guide

SUMMARY:
The purpose of this study is to present a guided lateral window sinus lift (GLSL) procedure with the aid of a fully digital workflow using surgical templates for window osteotomy preparation and implant placement.

DETAILED DESCRIPTION:
In Group 1; The surgical procedure began with the adaptation of a prefabricated guide to the surgical site, ensuring firm stabilization. Implant positions were marked, and after the removal of the guide, a crestal incision was made. A mucoperiosteal flap was reflected, exposing the maxillary sinus and alveolar crest. The guide was readapted, marking implant positions, and a lateral window was formed using a bur or piezotome. Sinus membrane elevation was performed carefully. Implants were placed with graft material beneath the elevated membrane. In cases of bony plate preservation, the window was covered. In Group 2 (Lateral Maxillary Sinus Floor Elevation without a surgical guide), a crestal incision and mucoperiosteal flap exposed the sinus. A bony window was created, and careful elevation of the sinus floor followed. Implant osteotomies were completed, and graft material was packed into the sinus. A resorbable membrane was applied, and the flap was sutured. NanoboneÒ was used as the standard graft material in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients (over 18 years of age), without any systemic complication.
* Patients who need for dental implant in posterior maxilla with bone height below the maxillary sinus is < 6 mm.
* Non smokers or patients who smoked less than 11 cig/day Will be included.

Exclusion Criteria:

* Uncontrolled systemic diseases which affect bone healing.
* Presence of any pathology in the site of operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Maxillary sinus volume | Preoperative, Immediate postoperative, 6 Months
  In cubic centimetre (cm3)

SECONDARY OUTCOMES:
Bone Gain | Immediate postoperative, 6 Months
  Im Millimeter (mm)
Implant stability | Intra-operative, 6 Months
  In implant stability quotient (ISQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR